CLINICAL TRIAL: NCT02669615
Title: A Phase II, Open-Label, Pharmacokinetic Study of Propylene Glycol-Free Melphalan HCl for Myeloablative Conditioning in Multiple Myeloma Patients Undergoing Autologous Transplantation
Brief Title: Pharmacokinetic Study of Propylene Glycol-Free Melphalan HCl for Myeloablative Conditioning in Multiple Myeloma Patients Undergoing Autologous Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Parameswaran Hari, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00026736
Record Dates: First submitted 2016-01-24; First posted 2016-02-01 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Melphalan HCl; Autologous Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Melphalan HCl for injection (propylene glycol free) (Experimental): Patients will receive 200 mg/m^2 of Melphalan HCl for injection (propylene glycol free) as a one-time infusion on day 2. Blood samples for the pharmacokinetic (PK) evaluation of melphalan will be collected after melphalan dosing (day -2). Following one day of rest after the myeloablative Melphalan conditioning (day -1), patients will receive an autologous graft with a minimum cell dose of 2 × 106 CD34+ cells/kg of patient body weight (day 0).
  Interventions: Drug: Melphalan HCl for injection (propylene glycol free)

INTERVENTIONS:
Drug: Melphalan HCl for injection (propylene glycol free) — During the study period, patients will receive 200 mg/m^2 of Melphalan HCl for injection (propylene glycol free) as a one-time infusion on day 2.

SUMMARY:
This study is a single-center, open-label study of high-dose Melphalan HCl (hydrochloric acid) for injection (propylene glycol-free Melphalan) conducted in 24 patients, who have symptomatic multiple myeloma and qualify for autologous stem-cell transplantation (ASCT).

There will be three distinct evaluation periods in this trial: a pretreatment period, a study period and a follow-up period.

DETAILED DESCRIPTION:
OVERVIEW: This study is a single-center, open-label study of high-dose Melphalan HCl for injection (propylene glycol free Melphalan) conducted in 24 patients, who have symptomatic multiple myeloma and qualify for ASCT.

There will be three distinct evaluation periods in this trial: a pretreatment period, a study period and a follow-up period.

PRETREATMENT:

Pretreatment Period Evaluations (Days -30 to -3). Baseline assessments will be collected within 30 days of dosing with Melphalan HCl for injection (propylene glycol free), after the patient has signed the informed consent. These include clinical and laboratory assessments (e.g., medical history and physical examination, hematology, urine analysis, creatinine clearance), chest X-ray and vital signs.

STUDY TREATMENT:

1. During the study period, patients will receive 200 mg/m^2 of Melphalan HCl for injection (propylene glycol free) as a one-time infusion on day
2. Following one day of rest after the myeloablative Melphalan conditioning (day -1), patients will receive an autologous graft with a minimum cell dose of 2 × 106 CD34+ cells/kg of patient body weight (day 0).
3. Pharmacokinetic, efficacy and safety evaluations will be performed during the study period.

FOLLOW-UP:

ASCT Day +1 until Day+100. During the follow-up period, patients will return for daily laboratory tests (hematology and basic serum chemistry) and will be evaluated weekly by their physicians until the engraftment date, with the final end-of-study evaluation occurring up to seven days after engraftment date. During the follow-up period, the tests (e.g., physical examination, CBC, vital signs, full serum chemistry panel, bone marrow biopsy) will be performed weekly until engraftment (unless otherwise specified).

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic multiple myeloma (MM) requiring treatment at or following diagnosis.
* Patients with MM, who qualify for ASCT therapy, and have received pretransplant therapy prior to transplantation.
* Adult patients (≥18 years of age) meeting local institutional criteria to receive a total Melphalan dose of 200 mg/m^2 as a conditioning regimen.
* Patients with an adequate autologous graft, which is defined as an unmanipulated, cryopreserved, peripheral blood cell graft containing at least 2 × 106 CD34+ cells/kg, based on patient weight.
* Patients with adequate organ function, as measured by:
* Cardiac: Left ventricular ejection fraction at rest >40% (documented within 30 days prior to Day -3).
* Hepatic: Bilirubin <2 × the upper limit of normal (ULN) and Alanine transaminase/Aspartate transaminase (ALT/AST) <3 × ULN.
* Renal: Creatinine clearance >40 mL/min (measured or calculated/estimated).
* Pulmonary: Adjusted Diffusing capacity of the lungs for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), forced vital capacity (FVC) >50% of predicted value (corrected for hemoglobin level [Hgb]) and documented within prior to day -3.

Exclusion Criteria:

* Patients with systemic AL amyloidosis (immunoglobulin light chain amyloidosis).
* Eastern Cooperative Oncology Group (ECOG) performance status ≥2.
* Patients with uncontrolled hypertension.
* Patients with a serious active bacterial, viral or fungal infection.
* Patients with prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent >5 years previously will be allowed. Cancer treated with curative intent <5 years previously will not be allowed unless approved by the medical monitor.
* Female patients who are pregnant (positive human chorionic gonadotropin [ß-HCG]) or breastfeeding.
* Female patients of childbearing potential, who are unwilling to use adequate contraceptive techniques during and for one month following study treatment with Melphalan HCl for injection (propylene glycol free).
* Patients seropositive for HIV.
* Patients who are unwilling to provide informed consent.
* Patients receiving other concurrent anticancer therapy (including chemotherapy, radiation, hormonal treatment, or immunotherapy, but excluding corticosteroids) within 30 days prior to the ASCT or planning to receive any of these treatments prior to study discharge.
* Patients concurrently participating in any other clinical study.
* Patients who are hypersensitive or intolerant to any component of the study drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Hari, MD, MRCP, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Melphalan HCl for Injection (Propylene Glycol Free): Patients will receive 200 mg/m^2 of Melphalan HCl for injection (propylene glycol free) as a one-time infusion on day 2. Blood samples for the pharmacokinetic (PK) evaluation of melphalan will be collected after melphalan dosing (day -2). Following one day of rest after the myeloablative Melphalan conditioning (day -1), patients will receive an autologous graft with a minimum cell dose of 2 × 106 CD34+ cells/kg of patient body weight (day 0).
  Melphalan HCl for injection (propylene glycol free): During the study period, patients will receive 200 mg/m2 of Melphalan HCl for injection (propylene glycol free) as a one-time infusion on day 2.
Period: Overall Study
Arm/Group | Melphalan HCl for Injection (Propylene Glycol Free)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Melphalan HCl for Injection (Propylene Glycol Free): Patients will receive 200 mg/m2 of Melphalan HCl for injection (propylene glycol free) as a one-time infusion on day 2. Blood samples for the pharmacokinetic (PK) evaluation of melphalan will be collected after melphalan dosing (day -2). Following one day of rest after the myeloablative Melphalan conditioning (day -1), patients will receive an autologous graft with a minimum cell dose of 2 × 106 CD34+ cells/kg of patient body weight (day 0).
  Melphalan HCl for injection (propylene glycol free): During the study period, patients will receive 200 mg/m2 of Melphalan HCl for injection (propylene glycol free) as a one-time infusion on day 2.
Arm/Group | Melphalan HCl for Injection (Propylene Glycol Free)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Pharmacokinetics)
Description: Maximum observed plasma concentration. Derived from the individual raw data.
Time Frame: Day -2
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Melphalan HCl for Injection (Propylene Glycol Free)
Number analyzed (Participants) | 24
ng/ml | 7380 [5220 to 11200]

2. Primary Outcome: AUC0-t (Pharmacokinetics)
Description: Area under the plasma concentration-time curve to the last measurable time point (AUC0-t) calculated by the trapezoidal rule. The area under the concentration-time curve (AUC) is calculated to determine the total drug exposure over a period of time.
Time Frame: Day -2
Measure: Median (Full Range); unit: ng*min/ml
Arm/Group | Melphalan HCl for Injection (Propylene Glycol Free)
Number analyzed (Participants) | 24
ng*min/ml | 533552 [253780 to 770538]

3. Secondary Outcome: Transplant-Related Mortality (TRM) Following Autologous Stem-Cell Transplantation (ASCT)
Description: TRM will be summarized descriptively (death within 100 days without relapse following ASCT).
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Melphalan HCl for Injection (Propylene Glycol Free)
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: 100 days post transplant
Arm/Group | Melphalan HCl for Injection (Propylene Glycol Free)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 24/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan HCl for Injection (Propylene Glycol Free) (N=24)
leukopenia (Blood and lymphatic system disorders) | 24 (24) — Myeloablation as expected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02669615/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02669615/SAP_001.pdf